CLINICAL TRIAL: NCT04525066
Title: Injection Thyroplasty During Transoral Laser Microsurgery for Early Glottic Cancer: Single-blinded Randomized Controlled Trial
Brief Title: Phonosurgical Augmentation After Laser Resection of Early Glottic Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ayhman Al Afif (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Ayhman Al Afif, Principal Investigator, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1020322
Record Dates: First submitted 2020-08-11; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Head and Neck Neoplasms; Head and Neck Squamous Cell Carcinoma; Voice Disorders; Laryngeal Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Voice Disorders; Laryngeal Neoplasms | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group - Receiving Hyaluronic Acid Injection (Experimental): Randomized group of patients receiving hyaluronic acid injection into the glottis during transoral laser microsurgery for early glottic cancer.
  Interventions: Drug: Hyaluronic acid
- Control Group - Not Receiving Hyaluronic Acid Injection (Placebo Comparator): Randomized group of patients not receiving hyaluronic acid injection into the glottis during transoral laser microsurgery for early glottic cancer.
  Interventions: Other: No Hyaluronic Acid Injection Injection

INTERVENTIONS:
Drug: Hyaluronic acid — Patients in the treatment group received hyaluronic acid injection into the unaffected vocal cord intra-operatively during transoral laser microsurgery for early glottic cancer.
  Other Names: Hyaluronic Acid Laryngoplasty
  Arms: Treatment Group - Receiving Hyaluronic Acid Injection
Other: No Hyaluronic Acid Injection Injection — Patients in the placebo group did not receive hyaluronic acid injection into the unaffected vocal cord intra-operatively during transoral laser microsurgery for early glottic cancer.
  Arms: Control Group - Not Receiving Hyaluronic Acid Injection

SUMMARY:
Objectives: Transoral Laser Microsurgery (TLM) is widely used in for treating T1/T2 glottic cancers. Hyaluronic acid (HA) is a safe and commonly-used injectable in vocal cord augmentation. We report on the results of our single-blinded, randomized-controlled trial (RCT) investigating the impact of intra-operative HA injection on voice outcomes in early glottic cancer.

Methods: Patients with T1/T2 glottic cancers were randomized to the treatment group (n=14) receiving HA injection to the unaffected cord during TLM; or the control group, receiving no injection (n=16). All patients had a Voice Handicap Index-10 (VHI-10) questionnaire and a Maximum Phonation Time (MPT) measurement preoperatively and at 3, 12 and 24 months post-operatively. Mean change in VHI-10 and MPT, between pre-operative and post-operative time points, and between the time points, were compared. Survival estimates were also calculated.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* 18 years of age or older with a biopsy-proven T1a, T1b or T2 glottic SCC
* Lesion amenable to CO2 TLM resection.

Exclusion Criteria:

* Previous radiotherapy to the head and neck.
* Palpable, or radiographic, pathological lymphadenopathy.
* Allergy, or sensitivity, to HA or components of the injectable.
* Neurological disorder affecting phonation, such as multiple sclerosis or stroke.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-08-13 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
Voice Outcome | Change at 3 months post-operatively compared to baseline.
  Voice Handicap Index-10 Scores
Voice Outcome | Changes at 12 months post-operatively compared to baseline.
  Voice Handicap Index-10 Scores
Voice Outcome | Changes at 24 months post-operatively compared to baseline.
  Voice Handicap Index-10 Scores
Voice Outcome | Changes at 3 months post-operatively compared to baseline.
  Maximum Phonation Time
Voice Outcome | Changes at 12 months post-operatively compared to baseline.
  Maximum Phonation Time
Voice Outcome | Changes at 24 months post-operatively compared to baseline.
  Maximum Phonation Time

SECONDARY OUTCOMES:
Overall survival | 24 months post-augmentation
  Kaplan-Meier Survival Analysis
Disease free survival | 24 months post-augmentation
  Kaplan-Meier Survival Analysis
Recurrence-free survival | 24 months post-augmentation
  Kaplan-Meier Survival Analysis

IPD SHARING:
Plan to Share IPD: No